CLINICAL TRIAL: NCT01175174
Title: Clinical, Airway Inflammatory, and HRA Phenotypes, in Preschool Children With Acute Asthmatic Attack Presenting to the ED.
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Avigdor Mandelberg, Director, Pediatric Pulmonry Unit, Wolfson Medical Center
Other Study IDs: 1038-sputum
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Asthma
Keywords: asthma; preschool children; adenosine provocation test; metacholine provocation test; pediatric emergency department
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical, Airway Inflammatory, and HRA Phenotypes, in preschool children with acute asthmatic attack presenting to the ED.

Background:

Children under the age of 5 years have the highest hospitalization rate of asthma. The most common causes of acute exacerbations of asthma requiring urgent medical care are viral respiratory infections. Most of these children < 6 y old are not atopic.

The inflammatory response to these mostly viral-induced asthmatic attacks is not well characterized in the literature. Moreover it is not known whether different kind of inflammatory responses exist in this population and how this correlate to clinical outcomes and clinical phenotypes in preschool children presenting ti the ED with acute asthmatic attack.

Therefore, the purpose of the present study is to:

Investigate the characterization of induced sputum cytology in preschool children with acute asthmatic attack and whether there is correlation between specific sputum cytology and response to therapy and to investigate airways hyper-responsiveness to adenosine 5'-monophosphate and to metacholine in pre school children 2-6 y old at 2 weeks and at 3 month following acute asthmatic exacerbation and look for correlation with response to treatment and sputum cytology. Clinical phenotypes of this patient population will also be investigated.

DETAILED DESCRIPTION:
Clinical, Airway Inflammatory, and HRA Phenotypes, in preschool children with acute asthmatic attack presenting to the ED.

Background:

Children under the age of 5 years have the highest hospitalization rate of asthma. The most common causes of acute exacerbations of asthma requiring urgent medical care are viral respiratory infections. Most of these children < 6 y old are not atopic.

The inflammatory response to these mostly viral-induced asthmatic attacks is not well characterized in the literature. Moreover it is not known whether different kind of inflammatory responses exist in this population and how this correlate to clinical outcomes and clinical phenotypes.

Therefore, the purpose of the present study is to:

Investigate the characterization of induced sputum cytology, bronchial hyper-responsiveness (BHR, and clinical phenotypes in preschool children with acute asthmatic attack presenting to the ED and whether there is correlation between specific sputum cytology and response to therapy.

and to investigate airways hyper-responsiveness (BHR)to adenosine 5'-monophosphate and to metacholine in pre school children 2-6 y old at 2 weeks and at 3 month following acute asthmatic exacerbation and look for correlation with response to treatment and sputum cytology.

Clinical phenotypes of this patient population will also be investigated.Clinical characteristics of the preschool children presenting to the ED with asthmatic attack will be compared to normal controls recruited from ambulatory clinics at the same area.

ELIGIBILITY:
Inclusion Criteria:

* children, age: 1-6 years old
* presenting to the ER with acute wheezing episode.

Exclusion Criteria:

* Any chronic (lung, cardiac, immunologic, neurologic) disease

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, age: 1-6 years old presenting to the emergency room (ER) with acute wheezing episode.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
airways inflammatory phenotype | Within 24 hours from admission to the emergency department (ED)
post attack bronchial hyperreactivity to adenosine 5'-monophosphate and to metacholine | 1. Within 2 weeks of recruitment 2. After 3 moths from recruitment

SECONDARY OUTCOMES:
Relationship between post attack bronchial hyperreactivity to adenosine 5'-monophosphate and to metacholine and the response to treatment and cytologic phenotypes. | 1. Within 3 weeks of recruitment 2. Beyond 3 moths from recruitment
relationship between cytologic phenotypes and response to treatment. | Within 3 months of recruitmant
clinical phenotype | whithin 1 month of presentation
  Clinical characteristics of the preschool children presenting to the ED with asthmatic attack will be compared to mormal controls recruited from ambulatory clinics at the same area.

CONTACTS AND LOCATIONS:
Overall Officials: Avigdor Mandelberg, MD, Study Chair — The Sackler School of Medicine, Tel Aviv University, Israel
Locations (1):
- The Edith Wlofson Medical Center, Holon, Israel